CLINICAL TRIAL: NCT01225302
Title: A Phase 1 Study of Linifanib (ABT-869) in Combination With Carboplatin/Paclitaxel in Japanese Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) as First-Line Treatment
Brief Title: A Study of Linifanib (ABT-869) in Combination With Carboplatin/Paclitaxel in Japanese Subjects With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W12-076
Record Dates: First submitted 2010-09-28; First posted 2010-10-21 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2012-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — linifanib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Linifanib; Drug: Carboplatin; Drug: Paclitaxel
- Arm B (Experimental)
  Interventions: Drug: Linifanib; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Linifanib — Low dose linifanib (once a day)
  Other Names: ABT-869
  Arms: Arm A
Drug: Linifanib — High dose linifanib (once a day)
  Other Names: ABT-869
  Arms: Arm B
Drug: Carboplatin — Given on Day 1 of every 21-day cycle
  Other Names: Paraplatin
Drug: Paclitaxel — Given on Day 1 of every 21-day cycle
  Other Names: Taxol

SUMMARY:
The primary objective of this study is to assess the safety and pharmacokinetics of linifanib, and identify tolerable dose of linifanib (ABT-869) in combination with carboplatin and paclitaxel in Japanese subjects with advanced or metastatic non-small cell lung cancer (NSCLC). Secondary objective is to obtain a preliminary efficacy of anti-tumor activity in the subjects as first-line treatment.

ELIGIBILITY:
Inclusion Criteria

* The subject must be 20 and older years of age.
* The subject must have cytologically or histologically confirmed non-squamous NSCLC. Subjects may have a mixed histology but must be predominantly non-squamous to be eligible.
* The subject must have advanced or metastatic (Stage IV [According to American Joint Committee on Cancer (AJCC) staging manual, 7th edition]) disease that is not amenable to surgical resection or radiation with curative intent.
* The subject must have not received prior chemotherapy for NSCLC.
* The subject has measurable disease, defined as at least 1 unidimensionally measurable lesion on a CT scan as defined by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
* The subject has an Easter Cooperative Oncology Group (ECOG) Performance Score of 0-1.
* The subject must have adequate bone marrow, renal and hepatic function.

Exclusion Criteria

* The subject has hypersensitivity to paclitaxel or to other drugs formulated with polyethoxylated castor oil (Cremophor).
* The subject has received any anti-cancer therapy for treatment of NSCLC including investigational agents, immunotherapy, traditional Chinese medicine/herbal remedies, hormonal, "targeted" agents (i.e., erlotinib, imatinib), biologic therapy or cytotoxic chemotherapy (i.e., alkylating agents, microtubule inhibitors, antimetabolites).
* The subject has a history of another active cancer within the past 5 years except cervical cancer in situ, in situ carcinoma of the bladder, squamous cell or basal cell carcinoma of the skin.
* The subject has active ulcerative colitis, Crohn's disease, celiac disease or any other conditions that interfere with absorption.
* The subject has a medical condition, which in the opinion of the study investigator places them at an unacceptably high risk for toxicities.
* The subject is pregnant or breast feeding.
* The subject has NSCLC with a predominant squamous cell histology.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety (Number of patients with adverse events and/or dose-limiting toxicities) | At each treatment visit (weekly for 6 weeks, then every 3 weeks)
  Evaluation of vital signs, physical exams, clinical lab testing and adverse event monitoring.

SECONDARY OUTCOMES:
Preliminary tumor response | Week 6
  Computed Tomography (CT) scan
Preliminary tumor response | Week 12
  Computed Tomography (CT) scan
Preliminary tumor response | Week 18
  Computed Tomography (CT) scan
Preliminary tumor response | Week 24
  Computed Tomography (CT) scan
Preliminary tumor response | Week 30
  Computed Tomography (CT) scan
Preliminary tumor response | Week 36
  Computed Tomography (CT) scan
Preliminary tumor response | Week 42
  Computed Tomography (CT) scan
Preliminary tumor response | Week 48
  Computed Tomography (CT) scan
Preliminary tumor response | Week 54
  Computed Tomography (CT) scan

CONTACTS AND LOCATIONS:
Overall Officials: Susumu Matsuki, BS, Study Director — Abbott Japan Co.,Ltd

REFERENCES:
- [Result] Horinouchi H, Yamamoto N, Nokihara H, Horai T, Nishio M, Ohyanagi F, Horiike A, Nakagawa K, Terashima M, Okabe T, Kaneda H, McKee MD, Carlson DM, Xiong H, Tamura T. A phase 1 study of linifanib in combination with carboplatin/paclitaxel as first-line treatment of Japanese patients with advanced or metastatic non-small cell lung cancer (NSCLC). Cancer Chemother Pharmacol. 2014 Jul;74(1):37-43. doi: 10.1007/s00280-014-2478-9. Epub 2014 May 8. PMID 24807459